CLINICAL TRIAL: NCT03479229
Title: Viveve Geneveve Treatment of the Vaginal Introitus to Evaluate Safety and Efficacy
Acronym: VIVEVE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viveve Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIVEVE II (VI-15-01)
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Female Sexual Dysfunction
Keywords: vaginal laxity; sexual function; vaginal childbirth; sexual dysfunction; diminished sexual function; satisfaction; arousal; desire; lubrication; orgasm
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Personal Satisfaction; Orgasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Geneveve Treatment (Experimental): Active Treatment
  Interventions: Device: Geneveve Treatment
- Sham Treatment (Placebo Comparator): Sham Treatment
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Geneveve Treatment — The active treatment group will receive a treatment dose of 90 J/cm^2
  Other Names: Active Treatment
  Arms: Geneveve Treatment
Device: Sham Treatment — The sham group will receive a sub-therapeutic dose of ≤ 1 J/cm^2.
  Arms: Sham Treatment

SUMMARY:
This study is evaluating the safety and efficacy of the Geneveve Treatment for women experiencing diminished sexual function following vaginal childbirth. Participants will be randomized to either active or sham treatment and followed for 12 months.

DETAILED DESCRIPTION:
Decreased sensation and decreased sexual satisfaction following vaginal childbirth has the potential to negatively impact overall sexual function and quality of life in many women. Previous research by obstetricians and gynecologists (OB/GYNs) found that changes in sexual health post-childbirth are not often discussed between physicians and their patients. One possible reason these discussions are not being initiated by physicians is the lack of an evidence-based treatment other than surgery.

While traditional surgery can be performed to improve sexual function following childbirth, pain at incision lines and scarring can lead to dyspareunia for months following the procedure, and a surgical procedure can be painful and the sutures may cause dense scarring. The post-operative recovery may last up to seven days before a woman can return to work. Resuming intercourse is not recommended for at least six weeks after these invasive surgeries. For the many women who are not good surgical candidates, due to health issues or situational limitations on downtime or their unwillingness to undergo a surgical procedure to improve sexual function, there is no other option.

The Geneveve Treatment offers a simple alternative to traditional surgery using non-ablative radiofrequency (RF) energy as a non-surgical approach to improve sexual function following vaginal childbirth. It induces a mild, controlled reaction in the submucosal tissues that stimulates the body to deposit collagen, thereby remodeling the tissue without causing scarring.

This study is designed to demonstrate that active treatment (i.e., Geneveve Treatment) is superior to the sham treatment for the primary efficacy and safety endpoints.

The active treatment group will receive a treatment dose of 90 J/cm^2 and the sham group will receive a sub-therapeutic dose of ≤ 1 J/cm^2. The participant, the investigator, and all study personnel will be blinded to the assignment for the entire study duration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at time of screening and pre-menopausal
* At least one vaginal delivery (> 37 completed weeks gestation)
* Sexual dysfunction
* Negative pregnancy test at Screening visit
* Sexually active

Exclusion Criteria:

* Currently breastfeeding or recently discontinued breastfeeding
* Medical history of keloid formation, genital fistula, thin recto-vaginal septum or obstetric trauma
* Implantable electrical device
* Medical or immunological condition
* Chronic use of anti-inflammatory drugs
* Current or previous use of local vaginal hormones
* Undergone previous elective surgical or non-invasive procedure(s) at the vaginal introitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) Total Score | 6 months post-treatment
  The FSFI is a 19-item validated measure of female sexual function. The FSFI consists of six domains: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. The recall period is the past 4 weeks. Each item's score can range from 0-5 (or 1-5 in several instances). For individual domain scores, the scores of the individual items that comprise the domain are summed, and the sum is multiplied by the domain factor. The six domain scores are summed to obtain the full scale score. It should be noted that within the individual domains, a domain score of zero indicates that the subject reported having no sexual activity during the past month. The total score is the sum of the domain scores and ranges from 2-36.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months post-treatment
  Safety as reported through Adverse Events from the time the subject signs the consent form through study completion.
Female Sexual Function Index (FSFI) Arousal Domain Score | 6 months post-treatment
  The FSFI is a 19-item validated measure of female sexual function. The FSFI Arousal domain recall period is the past 4 weeks. Each item's score can range from 0-5 (or 1-5 in several instances). For individual domain scores, the scores of the individual items that comprise the domain are summed, and the sum is multiplied by the domain factor. It should be noted that within the individual domains, a domain score of zero indicates that the subject reported having no sexual activity during the past month.
Female Sexual Function Index (FSFI) Orgasm Domain Score | 6 months post-treatment
  The FSFI is a 19-item validated measure of female sexual function. The FSFI Orgasm domain recall period is the past 4 weeks. Each item's score can range from 0-5 (or 1-5 in several instances). For individual domain scores, the scores of the individual items that comprise the domain are summed, and the sum is multiplied by the domain factor. It should be noted that within the individual domains, a domain score of zero indicates that the subject reported having no sexual activity during the past month.
Female Sexual Function Index (FSFI) Total Score | 12 months post-treatment
  The FSFI is a 19-item validated measure of female sexual function. The FSFI consists of six domains: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. The recall period is the past 4 weeks. Each item's score can range from 0-5 (or 1-5 in several instances). For individual domain scores, the scores of the individual items that comprise the domain are summed, and the sum is multiplied by the domain factor. The six domain scores are summed to obtain the full scale score. It should be noted that within the individual domains, a domain score of zero indicates that the subject reported having no sexual activity during the past month. The total score is the sum of the domain scores and ranges from 2-36.

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Bell, PhD, Study Director — Viveve Inc.
Locations (21):
- United States (19):
  - VIVEVE II Study Site, La Mesa, California
  - VIVEVE II Study Site, Orange, California
  - VIVEVE II Study Site, Denver, Colorado
  - VIVEVE II Study Site, Washington D.C., District of Columbia
  - VIVEVE II Study Site, Lake Worth, Florida
  - VIVEVE II Study Site, Plantation, Florida
  - VIVEVE II Study Site, West Palm Beach, Florida
  - VIVEVE II Study Site, Atlanta, Georgia
  - VIVEVE II Study Site, Idaho Falls, Idaho
  - VIVEVE II Study Site, Kalamazoo, Michigan
  - VIVEVE II Study Site, St Louis, Missouri
  - VIVEVE II Study Site, Omaha, Nebraska
  - VIVEVE II Study Site, New Brunswick, New Jersey
  - VIVEVE II Study Site, Albuquerque, New Mexico
  - VIVEVE II Study Site, New York, New York
  - VIVEVE II Study Site, Raleigh, North Carolina
  - VIVEVE II Study Site, Columbus, Ohio
  - VIVEVE II Study Site, Jackson, Tennessee
  - VIVEVE II Study Site, Tacoma, Washington
- Canada (2):
  - VIVEVE II Study Site, Calgary, Alberta
  - VIVEVE II Study Site, St. Johns, New Foundland